CLINICAL TRIAL: NCT06218784
Title: A Randomized, Double-blind, Placebo-controlled, Multiple-Ascending Dose Phase 1b Study to Evaluate the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Properties of iN1011-N17 After Oral Administration in Healthy Volunteers and Post-Herpetic Neuralgia Patients and to Assess the Relative Bioavailability of Mesylate vs Hydrochloride Salt Capsules in Healthy Volunteers
Brief Title: A MAD Study to Evaluate the Safety, Tolerability and PK/PD of iN1011-N17 in Healthy Volunteers and PHN Patients.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iN Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: iN1011-N17102
Record Dates: First submitted 2023-12-20; First posted 2024-01-23 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Post Herpetic Neuralgia; Pain; Osteoarthritis; Neuropathic Pain; Chronic Pain; Dorsal Root Ganglion; Nav 1.7
Keywords: Nav 1.7; Nav 1.7 inhibitor; Postoperative pain; Chemotherapy-induced neuropathic pain; Pain; Neurological Pain; Sodium Channel; Action Potential; Voltage Gated Sodium Channel; DRG Voltage Gated Sodium Channel 1.7; Sodium Channel 1.7; Volatage Gated Sodium Channel 1.7
MeSH Terms: conditions — Neuralgia, Postherpetic; Pain; Osteoarthritis; Neuralgia; Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- iN1011-N17 HCl Suspension (Part 1) (Experimental): Oral, Preformulation Suspension, b.i.d, Multiple Ascending Dose (Day 1~ Day7)
  Part 1:
  Participants will receive either iN1011-N17 or placebo in a 3:1 ratio. From Day 1 to Day 6, participants will receive iN1011-N17 or placebo b.i.d in the morning and in the evening, with approximately 12 hours between the 2 daily doses, and receive the last dose on Day 7 in the morning.
  Interventions: Drug: iN1011-N17 HCl Suspension (Part 1)
- iN1011-N17 HCl Capsule (Part 1) (Experimental): Oral, Nano Suspension Powder Capsule, b.i.d, Multiple Ascending Dose (Day 1~ Day7)
  Part 1:
  Participants will receive either iN1011-N17 or placebo in a 3:1 ratio. From Day 1 to Day 6, participants will receive iN1011-N17 or placebo b.i.d in the morning and in the evening, with approximately 12 hours between the 2 daily doses, and receive the last dose on Day 7 in the morning.
  Interventions: Drug: iN1011-N17 HCl Capsule (Part 1)
- Placebo Capsule (Part 1) (Placebo Comparator): Oral, Placebo capsule, b.i.d, Multiple Ascending Dose (Day 1~ Day7)
  Part 1:
  Participants will receive either iN1011-N17 or placebo in a 3:1 ratio. From Day 1 to Day 6, participants will receive iN1011-N17 or placebo b.i.d in the morning and in the evening, with approximately 12 hours between the 2 daily doses, and receive the last dose on Day 7 in the morning.
  Interventions: Drug: Placebo Capsule (Part 1)
- iN1011-N17 HCl Capsule (Part 2) (Experimental): Oral, Nano Suspension Powder Capsule, Single dose
  Part 2:
  2-period, randomized, open-label, crossover bioavailability part. Participants will receive a single oral dose of each study treatment (HCl salt and Mesylate salt), one during each of the 2 inpatient periods, in a randomized sequence of administration. There will be a minimum washout period of 5 days between each dose of study treatment.
  Interventions: Drug: iN1011-N17 HCl Capsule (Part 2)
- iN1011-N17 Mesylate Capsule (Part 2) (Active Comparator): Oral, AA10 Capsule, Single dose
  Part 2:
  2-period, randomized, open-label, crossover bioavailability part. Participants will receive a single oral dose of each study treatment (HCl salt and Mesylate salt), one during each of the 2 inpatient periods, in a randomized sequence of administration. There will be a minimum washout period of 5 days between each dose of study treatment.
  Interventions: Drug: iN1011-N17 Mesylate Capsule (Part 2)
- iN1011-N17 HCl Capsule (Part 3) (Experimental): Oral, Nano Suspension Powder Capsule, b.i.d, Multiple dose (Day 1~ Day7)
  Part 3:
  2 cohorts with up to 8 healthy volunteers and 8 PHN patients who will be randomized in a ratio of 3:1 to receive iN1011-N17 or placebo.
  Each participant in both cohorts will receive oral doses of iN1011-N17/ placebo b.i.d from Day 1 to Day 13, with approximately 12 hours between the 2 daily doses, and receive the last dose on Day 14 in the morning.
  Interventions: Drug: iN1011-N17 HCl Capsule (Part 3)
- iN1011-N17 Mesylate Capsule (Part 3) (Placebo Comparator): Oral, AA10 Capsule, b.i.d, Multiple dose (Day 1~ Day14)
  Part 3:
  2 cohorts with up to 8 healthy volunteers and 8 PHN patients who will be randomized in a ratio of 3:1 to receive iN1011-N17 or placebo.
  Each participant in both cohorts will receive oral doses of iN1011-N17/ placebo b.i.d from Day 1 to Day 13, with approximately 12 hours between the 2 daily doses, and receive the last dose on Day 14 in the morning.
  Interventions: Drug: iN1011-N17 Mesylate Capsule (Part 3)
- Placebo Capsule (Part 3) (Experimental): Oral, Placebo capsule, b.i.d, Multiple dose (Day 1~ Day14)
  Part 3:
  2 cohorts with up to 8 healthy volunteers and 8 PHN patients who will be randomized in a ratio of 3:1 to receive iN1011-N17 or placebo.
  Each participant in both cohorts will receive oral doses of iN1011-N17/ placebo b.i.d from Day 1 to Day 13, with approximately 12 hours between the 2 daily doses, and receive the last dose on Day 14 in the morning.
  Interventions: Drug: Placebo Capsule (Part 3)

INTERVENTIONS:
Drug: iN1011-N17 HCl Suspension (Part 1) — Dose: 100 mg b.i.d for 7 days (Multiple Ascending Dose)
  Arms: iN1011-N17 HCl Suspension (Part 1)
Drug: iN1011-N17 HCl Capsule (Part 1) — Dose: 200, 400, 800 mg b.i.d for 7 days (Multiple Ascending Dose)
  Arms: iN1011-N17 HCl Capsule (Part 1)
Drug: Placebo Capsule (Part 1) — Dose: b.i.d for 7 days
  Arms: Placebo Capsule (Part 1)
Drug: iN1011-N17 HCl Capsule (Part 2) — Dose: 400 mg QD
  Arms: iN1011-N17 HCl Capsule (Part 2)
Drug: iN1011-N17 Mesylate Capsule (Part 2) — Dose: 400 mg QD
  Arms: iN1011-N17 Mesylate Capsule (Part 2)
Drug: iN1011-N17 HCl Capsule (Part 3) — Dose: 400 mg b.i.d for 14 days
  Arms: iN1011-N17 HCl Capsule (Part 3)
Drug: iN1011-N17 Mesylate Capsule (Part 3) — Dose: 400 mg b.i.d for 14 days
  Arms: iN1011-N17 Mesylate Capsule (Part 3)
Drug: Placebo Capsule (Part 3) — Dose: b.i.d for 14 days
  Arms: Placebo Capsule (Part 3)

SUMMARY:
This study is a 3-part, Double-blind, Randomized, Placebo-controlled, Multiple Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics/Pharmacodynamic properties of iN1011-N17 after Oral Administration in Healthy Volunteers and Post-Herpetic Neuralgia patients, and to assess the relative bioavailability of Mesylate vs Hydrochloride salt capsules of iN1011-N17 in Healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers

1. Healthy male and female adults, aged 18 to 55 years of age (inclusive) at the time of consent.
2. Body mass index (BMI = body weight (kg)/[height (m)]2) between 18 kg/m2 and 32 kg/m2 (inclusive) at the time of Screening, and a minimum weight of 45 kg (inclusive).
3. Clinically acceptable pulse rate, RR, and tympanic body temperature (pulse rate between 45 and 100 beats per minute [bpm]; SBP between 90 and 140 mmHg; DBP between 50 and 90 mmHg; RR between 12 and 22 breaths/min; tympanic body temperature between 35.5°C and 37.7°C at Screening and Day -1). Measurements are to be recorded after a minimum of 5 minutes of resting in sitting or supine position

   For Healthy Volunteers and Post-Herpetic Neuralgia Patients
4. Clinical laboratory values within normal range as specified by the testing laboratory at Screening and Day -1, unless deemed not clinically significant by the Investigator.
5. All participants (excluding those who are exclusively in same-sex relationships, who are postmenopausal or have an exclusive partner who is postmenopausal) must agree to use a highly effective method of contraception throughout the study and for at least 30 days for females or 90 days for males after the last dose of IP. Female participants must not be breastfeeding, lactating, or pregnant during the study period.

   Female participants are required to be on their chosen contraceptive for at least 7 days before dosing.

   Female participants, where their sole, male sexual partner is vasectomized, must provide a verbal confirmation of azoospermia (90 days following the procedure) which should be recorded in the source documents by the Investigator.

   The minimum timeframe for pre-dose vasectomy for male participants is ≥ 12 weeks, unless they are the sole sexual partner of a female participant as outlined above.

   Male participants who are sexually active must use a condom combined with use of a highly-effective method of contraception for the female partner (excluding those who have had a vasectomy or whose partner is postmenopausal). Confirmation of the female partner's contraceptive information must be provided verbally by the male participant and should be recorded in the source documents by the Investigator. The postmenopausal status of the female partner must be confirmed verbally by the male participant and should be recorded in the source documents by the Investigator.
6. Cognitively capable of understanding the provided information and able to fully comply with protocol requirements.
7. Written informed consent prior to the commencement of any study procedures.
8. Willing and able to perform the necessary visits to the investigational site/institution.
9. In good general health at the Investigator's discretion, with no significant medical history, and with no clinically significant abnormalities on physical examination at Screening and before the first dose of IP.

   Post-Herpetic Neuralgia Patients
10. Male and female adults aged 50 to 75 years of age (inclusive) at the time of consent.
11. Clinically acceptable blood pressure (BP), pulse rate, RR, and tympanic body temperature (SBP between 90 and 140 mmHg; DBP between 50 and 95 mmHg; pulse rate between 45 and 100 bpm; RR between 12 and 22 breaths/min; tympanic body temperature between 35.5°C and 37.7°C) at Screening and Day -1. Measurements are to be recorded after a minimum of 5 minutes of resting in sitting or supine position.
12. BMI (body weight (kg)/[height (m)]2) between 18 kg/m2 and 40 kg/m2 (inclusive) at the time of Screening, and a minimum weight of 45 kg (inclusive).
13. A diagnosis of neuropathic pain of PHN is confirmed when the pain for >3 months after the herpes zoster rash is healed, with the pain area of a continuous area of affected rash.
14. Douleur Neuropathique 4 (DN4) score ≥4 at Screening.

Exclusion Criteria:

For Healthy Volunteers and Post-Herpetic Neuralgia Patients

1. Presence or history of carcinoma, hepatic, renal, neurological, pulmonary (except for childhood asthma), endocrine, hematologic, cardiovascular, or genitourinary disease that, in the opinion of the Investigator, may affect the evaluation of the IP or place the participant at undue risk (except for conditions that are stable on medications).
2. Presence of any underlying physical or psychiatric condition (except for conditions that are stable on medications) that, in the opinion of the Investigator, would undermine participant compliance to protocol requirements.
3. Presence or history of gastrointestinal disease (e.g., peptic ulcer, gastritis, gastric cramp, gastroesophageal reflex disease, Crohn's disease) or history of gastrointestinal surgery (except simple appendectomy or herniorrhaphy) that may affect assessment of safety and PK characteristics of the IP.
4. Presence or history of central nervous system disease that may affect assessment of safety and PK characteristics of the IP.
5. Presence of herniated disc (inter-vertebral, cervical or both) or history of related disease that, in the opinion of the Investigator, may affect assessment of safety and PK characteristics of the IP.
6. History of hypersensitivity to iN1011-N17 or to any of its components.
7. History of allergy or sensitivity to sulfonamides, hay fever, asthma, eczema, food allergies and/or allergies to other medications. Participants with asymptomatic, untreated, seasonal allergies at the time of dosing may be considered for inclusion on a case-by-case basis- PI and Sponsor approval must be obtained prior to randomization.
8. Any abnormal 12-lead ECG findings at Screening and Day -1, deemed by the Investigator or designee to be clinically significant.
9. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C (HCV), or human immunodeficiency virus (HIV) at Screening.
10. Positive urine drug screen test (including methamphetamines, opiates, cocaine, cannabinoids, phencyclidine, benzodiazepines, barbiturates, methadone, tricyclic antidepressants, and amphetamines) or alcohol breath test at Screening and Day -1. Repeated tests will be allowed at the discretion of the Investigator for suspected false positives.
11. Any of the following laboratory abnormalities within 14 days of the first treatment day:

    * Platelet count < 100,000 cells/mm3
    * Total neutrophil count < 1500 cells/mm3
    * Serum creatinine ≥ 1.5 x upper limit of normal (ULN)
    * Alanine aminotransferase (ALT) > 3.0 x ULN
    * Aspartate aminotransferase (AST) > 3.0 x ULN
    * Alkaline phosphatase > 2.0 x ULN
    * Bilirubin > 1.5 x ULN
    * Temperature ≥ 38°C or any other evidence of an infection
12. Use of any prescription drugs (except the ones mentioned in Section 7.4.1) within 14 days, and over the counter (OTC) medications, herbal remedies (including St John's Wort), dietary supplements or vitamins within 7 days, or five half-lives of the product, whichever is longer, before the first dose of IP and for the duration of the study without prior approval of the Investigator and the MM. This includes analgesics such as paracetamol and non-steroidal anti-inflammatories (for healthy volunteers only).
13. The use of any IP or investigational medical device within 30 days prior to Screening, or five half-lives of the product, whichever is longer.
14. Blood or plasma donation of more than 450 mL within 90 days before the first dose of IP and for the duration of the study. It is recommended that blood/plasma donations not be made for at least 30 days after study completion.
15. History of alcoholism, substance or drug abuse-related disorders deemed significant by the Investigator (or designee) (i.e., participants consuming > 21 units of alcohol per week for males and > 14 units of alcohol per week for females in the 90 days prior to dosing will be excluded. One unit of alcohol equals ½ pint [285 mL] of beer or lager, 1 glass [125 mL] of wine, or 1/6 gill [25 mL] of spirits).
16. Use of more than 5 nicotine-based products (including smoking tobacco, smokeless tobacco, and nicotine patches) per week, within 90 days prior to Screening. Volunteers must have a negative urine cotinine test at both Screening and Day -1 and refrain from the use of any nicotine-based products for the duration of the study.
17. Consumption of beverages or foods that contain grapefruit, star fruit, pomelos, or products containing these fruits, from 7 days, or from the time that is deemed significant by the Investigator, and products containing caffeine (e.g., coffee, green tea, black tea, and sodas) from 48 hours before the first dose of IP until discharge from the study unit (includes the period between Periods 1 and 2 in Part 2).
18. Unwilling to refrain from strenuous exercise from 48 hours prior to admission to the investigational site/institution and for the duration of the study, where strenuous exercise is defined as that which requires significant effort, energy, or strength, such as lifting weights or running.
19. Any other reason that, in the opinion of the Investigator, may affect assessment of safety, PK, or PD characteristics of the IP.
20. Have previously completed or withdrawn from this study or any other study investigating iN1011-N17 or have previously received the IP (for healthy volunteers only).
21. Received an investigational vaccine within 6 months, a live attenuated vaccine within 60 days, or a registered vaccine within 14 days prior to the Day -1 (Baseline visit).

    Post-Herpetic Neuralgia Patients
22. PI-NRS score of PHN-associated neuropathic pain over the last 24 hours at randomization of ≥9 or at least a daily pain score of ≥9 during the Washout Period.
23. Previous use of neurolytic block (e.g. chemical neurolytic block using phenol or ethyl alcohol, or radiofrequency thermocoagulation) or neurosurgical therapy for current PHN.
24. Other severe pain or the presence of other skin diseases or pain at the site of the rash at Screening or randomization unrelated to PHN, that may confound the assessment of PHN.
25. Participants who are unable or unwilling to cease the use of all pain medications, prescription and otherwise, as of the first day of the study Washout Period and until after Day 14 of the study. This includes all lamotrigine, carbamazepine, oxcarbazepine, mexiletine, valproate, lidocaine, lacosamide, amitriptyline, topiramate, selegiline, rasagiline medications. This excludes the use of paracetamol provided that a participant is able and willing to utilize a maximum of 4 g of paracetamol per 24-hour period as of the first day of the study Washout Period and until after Day 14 of the study. Common and approved medications for PHN patients are permitted if part of a stable treatment regimen (please refer to Section 7.4.1 for a list of permitted medications).
26. Participants who are unable or unwilling to cease the use of prohibited medication (in Section 7.4.1) during the whole study period. Have previously received the IP or any other investigational drug/device within 30 days or 5 half-lives, whichever is greater.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-07-29 (Estimated); Study Completion 2024-07-29 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and causality of AEs and serious AEs (SAEs) | Part 1: From baseline until follow-up, an average of 14 days Part 2: From baseline until follow-up, an average of 22 days Part 3: From baseline until follow-up, up to 21 days
Incidence of Physical examination abnormalities | Part 1: From baseline until follow-up, an average of 14 days Part 2: From baseline until follow-up, an average of 22 days Part 3: From baseline until follow-up, up to 21 days
Incidence of Vital signs abnormalities | Part 1: From baseline until follow-up, an average of 14 days Part 2: From baseline until follow-up, an average of 22 days Part 3: From baseline until follow-up, up to 21 days
Incidence of 12-lead ECG abnormalities | Part 1: From baseline until follow-up, an average of 14 days Part 2: From baseline until follow-up, an average of 22 days Part 3: From baseline until follow-up, up to 21 days
Incidence of Continous cardiac telemetry abnormalities | Part 1: From baseline until follow-up, an average of 14 days Part 2: From baseline until follow-up, an average of 22 days Part 3: From baseline until follow-up, up to 21 days
Incidence of Laboratory tests abnormalities | Part 1: From baseline until follow-up, an average of 14 days Part 2: From baseline until follow-up, an average of 22 days Part 3: From baseline until follow-up, up to 21 days

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Part 1: Day 1 Part 2: 0-72 hours post dose Part 3: Day 1
Time to maximum plasma concentration (Tmax) | Part 1: Day 1 Part 2: 0-72 hours post dose Part 3: Day 1
Terminal half-life (t1/2) | Part 1: Day 1 Part 2: 0-72 hours post dose Part 3: Day 1
Area under the plasma concentration curve (AUC0-12, AUC0-t, AUCinf) | Part 1: Day 1 and Day 7 Part 2: 0-72 hours post dose Part 3: Day 1 and Day 14
Percentage of AUCinf based on extrapolation (AUC%extrap) | Part 1: Day 1 and Day 7 Part 2: 0-72 hours post dose Part 3: Day 1 and Day 14
Apparent volume of distribution (Vz/F) | Part 1: Day 1 and Day 7 Part 3: Day 1 and Day 14
Apparent plasma elimination rate constant (λz) | Part 1: Day 1 and Day 7 Part 3: Day 1
Apparent clearance (CL/F) | Part 1: Day 1 Part 3: Day 1
Fraction excreted unchanged in urine (fe) | Part 1: Day 1 and Day 7 Part 3: Day 1 and Day 14
Amount of drug excreted unchanged in the urine (Ae) | Part 1: Day 1 and Day 7 Part 3: Day 1 and Day 14
Renal clearance (CLR) | Part 1: Day 1 and Day 7 Part 3: Day 1 and Day 14
Mean residence time (MRT) | Part 1: Day 1 and Day 7 Part 3: Day 1 and Day 14
Maximum (peak) steady-state plasma drug concentration during a dosage interval (Cmax,ss) | Part 1: Day 7 Part 3: Day 14
Minimum steady-state plasma drug concentration during a dosage interval (Cmin,ss) | Part 1: Day 7 Part 3: Day 14
Average steady-state plasma drug concentration during multiple-dose administration (Cav,ss) | Part 1: Day 7 Part 3: Day 14
Time to reach maximum (peak) plasma concentration following drug administration at steady-state (Tmax,ss) | Part 1: Day 7 Part 3: Day 14
Area under the plasma concentration-time curve during a dosage interval (τ) (AUCτ) | Part 1: Day 7 Part 3: Day 14
Apparent clearance at steady state (CLss/F) | Part 1: Day 7 Part 3: Day 14
Apparent volume of distribution at steady state (Vz,ss/F) | Part 1: Day 7 Part 3: Day 14
Accumulation ratio of Cmax and AUC (RAcmax or RAAUC) | Part 1: Day 7 Part 3: Day 14

OTHER OUTCOMES:
Daily pain intensity is assessed using the Daily Pain Score (DPS), which is an 11-point numeric scale ranging from 0, indicating 'no pain', to 10, indicating 'pain as bad as you can imagine'. | From baseline to Day 21
  Part 3 PHN patients
Score of Short Form McGill Pain Questionnaire (SF-MPQ) (Consists of 11 items. Uses a 4-point numeric scale ranging from 0, indicating 'none', to 4, indicating 'severe'.) | From baseline to Day 21
  Part 3 PHN patients
Score of Brief Pain Inventory Short Form (BPI-SF). (measures pain intensity, its effect on functionality and impact of pain. Uses a 11-point numeric scale ranging from 0, indicating 'no pain', to 10, indicating 'pain as bad as you can imagine'.) | From baseline to Day 21
  Part 3 PHN patients
Change in DPS score from Baseline Days 4, 7, 10, 14 and 21, based on daily pain assessment. | From baseline to Day 21
  Part 3 PHN patients
Change from Baseline in parameters assessed using SF-MPQ. | From baseline to Day 21
  Part 3 PHN patients
Change from Baseline in parameters assessed using BPI-SF (measurements of pain intensity, functionality, and impact of pain). | From baseline to Day 21
  Part 3 PHN patients
Proportion of patients experiencing a ≥ 30% decrease (improvement) in pain | From baseline to Day 21
  Part 3 PHN patients The scoring will be based on the daily pain intensity score (DPS), which is an 11-point numeric scale ranging from 0 to 10.
Change from period baseline values (time, s) in Cold pressor test (PDT, PTT) | From baseline to Day 14
  Part 3 healthy volunteers
Change from period baseline values (temperature, ℃) in Capsaicin 1% cream test (PDT, PTT) | From baseline to Day 14
  Part 3 healthy volunteers
Incidence of abnormalities: Thermal detection thresholds for the perception of cold and heat (CDT, HDT) | Baseline, Day 1 and Day 14
  Part 1 and Part 3 healthy volunteers
Incidence of abnormalities: Thermal pain thresholds for cold and heat threshold stimuli (CPT, HPT) | Baseline, Day 1 and Day 14
  Part 1 and Part 3 healthy volunteers
Incidence of abnormalities: Mechanical detection threshold and mechanical pain threshold (MDT, MPT) | Baseline, Day 1 and Day 14
  Part 1 and Part 3 healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia